CLINICAL TRIAL: NCT03043677
Title: Ex-vivo Modulatory Effect of Biological Drugs for Inflammatory Bowel Disease on the Mucosa and on Peripheral Blood Mononuclear Cells
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Javier P. Gisbert, PhD, MD, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: JPG-VED-2016-01
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab; golimumab; Adalimumab; vedolizumab; Ustekinumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cell culture supernatants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-inflamed
  Interventions: Biological: Ex-vivo stimulation of cells with infliximab, golimumab, adalimumab, vedolizumab and ustekinumab
- Inflamed ulcerative colitis
  Interventions: Biological: Ex-vivo stimulation of cells with infliximab, golimumab, adalimumab, vedolizumab and ustekinumab
- inflamed Crohn´s disease
  Interventions: Biological: Ex-vivo stimulation of cells with infliximab, golimumab, adalimumab, vedolizumab and ustekinumab

INTERVENTIONS:
Biological: Ex-vivo stimulation of cells with infliximab, golimumab, adalimumab, vedolizumab and ustekinumab — Ex-vivo conditioning of lamina propria and peripheral blood mononuclear cells.
  Here, we will address whether the current available biological therapies for IBD patients (infliximab, golimumab, adalimumab, vedolizumab and ustekinumab) elicit a differential effect on the mucosal capacity to recruit circulating leukocytes on an ex-vivo approach using transwell culture systems.

SUMMARY:
To characterize circulating DC subsets from healthy controls and IBD patients and to assess, following an ex vivo challenge, the effect of anti-TNF (infliximab, adalimumab and golimumab), anti-p40 -IL-12/IL-23- (ustekinumab) and anti-α4β7 (vedolizumab) immunomodulators on both the GI production of soluble immune mediators and the mucosal capacity to alter the recruitment capacity of circulating DC subsets. It is expected that such approach will provide further information on the action mechanisms of such therapies on IBD patients, allowing a better understanding of the pathophysiology of this disease and the identification of tissue-specific therapeutic targets, thus avoiding collateral problems associated with systemic immunomodulation.

ELIGIBILITY:
Inclusion Criteria:

Patients with active IBD, and endoscopic and histological diagnosis of CD or UC that attend a colonoscopy with sedation performed by medical criteria.

Patients without an IBD diagnosis, or other types of inflammatory, allergic, malignant or autoimmune diseases, prior to their inclusion in this project. All patients will attend a colonoscopy with sedation at medical judgment with biopsy indication for histopathological study as in cases of diarrhea but also due to changes in the bowel transit, rectal bleeding or screening for gastrointestinal diseases. Patients will be paired in age and gender with the IBD groups. All patients will have no signs of macroscopic or microscopic inflammation hence excluding the presence of microscopic colitis.

Exclusion Criteria:

1. Age less than 18 years
2. Chronic disease or any other advanced clinically significant pathology, uncontrolled by investigator judgment.
3. Should be with medication, this will be unchanged in the 3 months prior to colonoscopy.
4. Alcohol or drugs.
5. Pregnancy or lactation
6. Do not sign the informed consent form (see "Ethical Issues") In any case NO colonoscopies exclusively targeted for sampling for this project will be made

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy controls and patients with active inflammatory bowel disease (ulcerative colitis and Crohn´s disease).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Effect of biological drugs on the secretion of gut-chemoattractants by the intestinal mucosa | 18 months
  To assess, ex-vivo, the capacity of the IBD mucosa to recruit subsets of circulating leukocytes following mucosal conditioning with biological drugs.

IPD SHARING:
Plan to Share IPD: No